CLINICAL TRIAL: NCT05557318
Title: Using Micro Electro Mechanical Systems to Detect the Air of Vaginal Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taiwan Carbon Nano Technology Corporation (Industry)
Collaborators: Ainos, Inc. (f/k/a Amarillo Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A202203003
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Vaginal Infection; Vaginitis
Keywords: E-Nose
MeSH Terms: conditions — Vaginitis | interventions — Reverse Transcriptase Polymerase Chain Reaction; Culture Techniques

STUDY DESIGN:
Intervention Model Description: This clinical study is a prospective study to evaluate the sensitivity and specificity of the Ainos Flora Female Vaginal Health Tester in identifying vaginal infections. Potential subjects will be patients in the gynecological clinic. The study will evaluate the performance of the Ainos Flora Female Vaginal Health Tester by comparing it to the conventional real-time polymerase chain reaction (RT-PCR) and culture methods for the diagnosis of vaginitis to calculate both sensitivity and specificity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bacterial infections (Experimental): The subject is infected with at least one of the following pathogens:
  Bacterial vaginosis (BV) / Escherichia coli / Trichomonas / Group B streptococcus / Chlamydia trachomatis / Neisseria gonorrhoeae
  Interventions: Device: Vaginal swab for RT-PCR; Device: Vaginal swab for culture; Device: Metabolic gas signatures detected by Ainos Flora (operated by participant); Device: Metabolic gas signatures detected by Ainos Flora (operated by medical staff)
- Fungal infection : (Experimental): The subject is infected with Candida albicans only.
  Interventions: Device: Vaginal swab for RT-PCR; Device: Vaginal swab for culture; Device: Metabolic gas signatures detected by Ainos Flora (operated by participant); Device: Metabolic gas signatures detected by Ainos Flora (operated by medical staff)
- Mixed infection (Experimental): Bacterial and fungal infections coexist.
  Interventions: Device: Vaginal swab for RT-PCR; Device: Vaginal swab for culture; Device: Metabolic gas signatures detected by Ainos Flora (operated by participant); Device: Metabolic gas signatures detected by Ainos Flora (operated by medical staff)
- No infection (Experimental): Healthy participant
  Interventions: Device: Vaginal swab for RT-PCR; Device: Vaginal swab for culture; Device: Metabolic gas signatures detected by Ainos Flora (operated by participant); Device: Metabolic gas signatures detected by Ainos Flora (operated by medical staff)

INTERVENTIONS:
Device: Vaginal swab for RT-PCR — Screening for Bacterial vaginosis (BV) / Trichomonas / Chlamydia trachomatis / Candida albicans
Device: Vaginal swab for culture — Screening for Group B streptococcus / Neisseria gonorrhoeae / Escherichia coli
Device: Metabolic gas signatures detected by Ainos Flora (operated by participant) — The participant operates the Ainos Flora to collect signatures of metabolic gases in the vagina by herself.
Device: Metabolic gas signatures detected by Ainos Flora (operated by medical staff) — The medical staff operates the Ainos Flora to collect signatures of metabolic gases in the participant's vagina.

SUMMARY:
This clinical study aims to train the algorithm and assess the performance of the Ainos Flora Women's Vaginal Health Tester in identifying vaginal infections.

DETAILED DESCRIPTION:
Ainos Flora Women's Vaginal Health Tester is an in vitro diagnostic device implementing electronic nose technology to detect vaginal infections by examining metabolized gases of vaginal bacteria. The electronic nose system mainly comprises the Micro-Electro-Mechanical Systems (MEMS) gas sensor array and the Artificial Neural Network algorithm. The primary purpose of this study is to train the algorithm and assess the performance of the Ainos Flora in identifying vaginal infections. In addition, the primary outcome measures of this study, including sensitivity and specificity, will be used as a reference for the feasibility and sample size assessment of the next phase of pivotal clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Female, Age ≥20 to ≤50.
* Have had sexual experience.
* Fully understand the subject's informed consent process and be willing to undergo all study-related assessments and procedures.

Exclusion Criteria:

Women who meet any of the following criteria by participant report will be excluded from the study:

* During menstruation.
* Have performed vaginal washing within three days.
* Have been treated for vaginal infections within one week.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 120 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To assess the sensitivity and specificity of Ainos Flora in subjects compared to RT-PCR and culture groups in identifying the types of vaginitis. | Up to 6 months.
  * Bacterial infection : Bacterial vaginosis (BV) / Escherichia coli / Trichomonas / Group B streptococcus / Chlamydia trachomatis / Neisseria gonorrhea
  * Fungal infection: Candida albicans
  * Mixed infection: Bacterial and fungal infections coexist
  * No infection: Healthy participant

SECONDARY OUTCOMES:
Assess the change in sensitivity as the number of subjects is changed. | Up to 6 months.
  When the number of subjects reaches 30,60,90,120, input the collected gas data into the algorithm and calculate the sensitivity. We can then assess the change in sensitivity when the number of subjects changes from 30 to 60, 90, and 120.
Assess the change in specificity as the number of subjects is changed. | Up to 6 months.
  When the number of subjects reaches 30,60,90,120, input the collected gas data into the algorithm and calculate the specificity. We can then assess the change in specificity when the number of subjects changes from 30 to 60, 90, and 120.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Fung-Wei Chang, Principal Investigator — Tri-Service General Hospital
Locations (2):
- Taiwan (2):
  - MacKay Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No